CLINICAL TRIAL: NCT05401409
Title: Double-Blind, Randomised Placebo-Controlled Study to Determine the Effect of Beetroot Juice on Reducing Blood Pressure in Hypertensive Adults With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Effect of Beetroot Juice on Reducing Hypertension in Autosomal Dominant Polycystic Kidney Disease
Acronym: BEET-PKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Collaborators: Westmead Institute for Medical Research (Unknown)
Responsible Party: Principal Investigator, Gopala K. Rangan, Nephrologist, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020_ETH01718
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Autosomal Dominant Polycystic Kidney; Hypertension; Endothelial Dysfunction
Keywords: Autosomal Dominant Polycystic Kidney Disease; ADPKD; Beetroot juice; Hypertension; Nitrate supplementation; Nitric oxide
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich beetroot juice (Experimental): Beetroot juice containing naturally occurring nitrate (400mg total nitrate)
  Interventions: Dietary Supplement: Beetroot juice
- Nitrate-depleted beetroot juice (Placebo Comparator): Beetroot juice with nitrate removed
  Interventions: Dietary Supplement: Nitrate-depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — 70mls beetroot juice (400mg nitrate) given daily for 4 weeks
  Other Names: Beet It Sport Shot
  Arms: Nitrate-rich beetroot juice
Dietary Supplement: Nitrate-depleted beetroot juice — 70mls beetroot juice (nitrate-depleted) given daily for 4 weeks
  Arms: Nitrate-depleted beetroot juice

SUMMARY:
People with autosomal dominant polycystic kidney disease (ADPKD) develop high blood pressure and kidney disease. Previous studies have shown that a commonly occurring chemical, nitric oxide (NO), is reduced in ADPKD, and may contribute, in part, to high blood pressure in this condition. Nitrate is found in high concentrations naturally in beetroots, and increases NO. The aim of this study is to determine if beetroot juice reduces blood pressure in hypertensive people with ADPKD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autosomal Dominant Polycystic Kidney Disease
* Age > 18 years old
* Estimated Glomerular Filtration Rate (eGFR) > 30 mL/min/1.73m2
* Treatment with at least one anti-hypertensive

Exclusion Criteria:

* Inability to provide Informed Consent
* Labile, unstable, uncontrolled hypertension and/or changes in BP treatment 28 days prior to the screening visit
* Non-compliance with study procedures and/or daily BP measurements during the screening period
* Medical conditions or treatments that might interfere with the generation of NO metabolites or the primary endpoint (e.g. nitrate drugs; cigarette smoking; unwilling to stop using antiseptic mouthwash; severe, uncontrolled hypercholesterolemia; pregnancy or post-partum and lactating)
* Any serious or other medical conditions that might interfere with follow-up or stability of blood pressure (e.g. current active malignancies; uncontrolled diabetes mellitus with elevated HbA1c > 10%)
* Dislike of taste of beetroot juice
* Allergy to beetroot
* Enrolled in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G K Rangan, Principal Investigator — Westmead Hospital, Western Sydney Local Health District
Locations (2):
- Australia (2):
  - Westmead Hospital, Sydney, New South Wales
  - Westmead Institute for Medical Research, Westmead, New South Wales

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Sagar PS, Munt A, Saravanabavan S, Vahedi FA, Elhindi J, Nguyen B, Chau K, Harris DC, Lee V, Sud K, Wong N, Rangan GK. Efficacy of beetroot juice on reducing blood pressure in hypertensive adults with autosomal dominant polycystic kidney disease (BEET-PKD): study protocol for a double-blind, randomised, placebo-controlled trial. Trials. 2023 Jul 29;24(1):482. doi: 10.1186/s13063-023-07519-2. PMID 37507763

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitrate-rich Beetroot Juice | Nitrate-depleted Beetroot Juice
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrate-rich Beetroot Juice | Nitrate-depleted Beetroot Juice | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.5) | 49.3 (12.46) | 49.4 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 17 | 16 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-reported ethnicity
  Participants
    Caucasian | 20 | 22 | 42
    Asian | 8 | 7 | 15
    Other | 2 | 1 | 3
Employment status, categorical (Part time, Full time)) [Count of Participants; unit: Participants]
  Full time | 22 | 26 | 48
  Part time | 7 | 4 | 11
  Umemployed | 1 | 0 | 1
Factor precipitating diagnosis, categorical (family history screening; pain; hypertension;incidental [Count of Participants; unit: Participants]
  Screening (family history) | 12 | 13 | 25
  Pain | 3 | 6 | 9
  Hypertension | 8 | 2 | 10
  Incidental | 2 | 5 | 7
  Other | 5 | 4 | 9
Diagnosis confirmatory test (radiographic) [Count of Participants; unit: Participants] | 30 | 30 | 60
Age at diagnosis [Mean (Standard Deviation); unit: years] | 30.9 (13.31) | 33.1 (13.1) | 32 (13.2)
Family history of ADPKD [Count of Participants; unit: Participants]
  Yes | 22 | 23 | 45
  No | 8 | 4 | 12
  Unknown | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinic Systolic and Diastolic Blood Pressure From Baseline to 4 Weeks (End of Study)
Description: Change in systolic and diastolic blood pressure over two time points - from readings taken at baseline (visit 1) compared with readings taken at 4 weeks (which was the end of the study; visit 3)
Time Frame: 4 weeks
Population: One patient in the nitrate-rich group was lost to follow-up.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nitrate-rich Beetroot Juice | Nitrate-depleted Beetroot Juice
Number analyzed (Participants) | 29 | 30
mmHg
  Systolic blood pressure | -5.36 (12.69) | -7.65 (14.07)
  Diastolic blood pressure | -3.55 (7.08) | -2.73 (7.81)

2. Secondary Outcome: Average Change in Daily Home Systolic and Diastolic Blood Pressure Per Week, Over 4 Weeks
Description: Reported change in blood pressure is average change per week, over 4 weeks
Time Frame: 4 weeks
Measure: Mean (95% Confidence Interval); unit: mmHg/week
Arm/Group | Nitrate-rich Beetroot Juice | Nitrate-depleted Beetroot Juice
Number analyzed (Participants) | 29 | 30
mmHg/week
  Systolic blood pressure | -0.51 [-1.40 to 0.38] | -0.55 [-1.42 to 0.31]
  Diastolic blood pressure | -0.24 [-0.85 to 0.38] | -0.47 [-1.07 to 0.13]

3. Secondary Outcome: Urinary Albumin to Creatinine Ratio at Baseline and at 4 Weeks (End of Study)
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: mg/mmol
Arm/Group | Nitrate-rich Beetroot Juice | Nitrate-depleted Beetroot Juice
Number analyzed (Participants) | 29 | 30
mg/mmol
  Baseline | 2.2 [0.4 to 5.4] | 3.9 [1.7 to 9.0]
  4 weeks (end of study) | 2.5 [0.2 to 5.8] | 3.6 [0.9 to 13.9]

4. Secondary Outcome: Change in Serum Nitric Oxide Metabolite Levels From Baseline to 4 Weeks (End of the Study)
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: µM
Arm/Group | Nitrate-rich Beetroot Juice | Nitrate-depleted Beetroot Juice
Number analyzed (Participants) | 29 | 30
µM | 20.08 [6.60 to 30.68] | 0.97 [-1.83 to 3.71]

5. Secondary Outcome: Change in Salivary Nitric Oxide Metabolite Levels From Baseline to 4 Weeks (End of the Study)
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2028-12

6. Secondary Outcome: Serum Asymmetric Dimethylarginine at Baseline and at 4 Weeks (End of the Study)
Description: Asymmetric dimethylarginine (ADMA) which is a recognized marker of endothelial dysfunction and inhibitor of nitric oxide
Time Frame: 4 weeks
Measure: Median (Standard Deviation); unit: umol/L
Arm/Group | Nitrate-rich Beetroot Juice | Nitrate-depleted Beetroot Juice
Number analyzed (Participants) | 29 | 30
umol/L
  Baseline ADMA level | 0.47 (0.08) | 0.47 (0.09)
  4 week ADMA level (end of study) | 0.50 (0.10) | 0.52 (0.11)

ADVERSE EVENTS:
Time Frame: 4 weeks (from enrollment to end of follow up)
Arm/Group | Nitrate-rich Beetroot Juice | Nitrate-depleted Beetroot Juice
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 18/29 | 11/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nitrate-rich Beetroot Juice (N=29) | Nitrate-depleted Beetroot Juice (N=30)
Gastrointestinal symptoms (not serious adverse event) (Gastrointestinal disorders) | 13 | 10
Change in bowel habit (Gastrointestinal disorders) | 12 | 8 — Includes all changes in bowel habit, including those perceived as positive changes
Bloating (Gastrointestinal disorders) | 5 | 2
Gastritis (Gastrointestinal disorders) | 1 | 3
Beeturia (Renal and urinary disorders) | 15 | 7
Beet-coloured faeces (Gastrointestinal disorders) | 18 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT05401409/Prot_SAP_000.pdf